CLINICAL TRIAL: NCT03700346
Title: Muscle Lactate and Lactate to Pyruvate Ratio Clearance as Useful Biomarkers for the Prediction of Mortality in Septic Shock Patients
Brief Title: Muscle Lactate and Lactate to Pyruvate Ratio Clearance in Septic Shock Patients
Acronym: ClMLsepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Military Hospital of Tunis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MilitaryHospTunis
Record Dates: First submitted 2018-09-30; First posted 2018-10-09 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Microdialysis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- survivors (Other): survivor at ICU discharge muscle microdialysis
  Interventions: Device: microdialysis
- Non survivors (Other): death before ICU discharge muscle microdialysis
  Interventions: Device: microdialysis

INTERVENTIONS:
Device: microdialysis — Interstitial tissue concentrations of lactate, pyruvate, glucose and glycerol were obtained by using muscle microdialysis

SUMMARY:
We conducted this study aiming to assess the performance of muscle Lactate and lactate to pyruvate (L/P) ratio clearance in predicting mortality in septic shock patients by using microdialysis.

DETAILED DESCRIPTION:
Microcirculatory alterations are frequently observed in patients with sepsis. In vivo microdialysis (MD) is a bedside technique that can monitor tissue metabolic changes. We conducted this study aiming to assess the performance of muscle Lactate and lactate to pyruvate (L/P) ratio clearance in predicting mortality in septic shock patients by using microdialysis.

Interstitial tissue concentrations of lactate, pyruvate, glucose and glycerol were obtained at baseline and every 6 hours for 3 days by using muscle microdialysis. Clearances of muscle lactate, and L/P ratio were defined as the percentage change in muscle lactate level or L/P ratio compared to baseline (H0) values. A positive value of clearance means a decrease in the rate of the parameter under study.

ELIGIBILITY:
Inclusion Criteria:

* patients fulfilled the criteria of septic shock

Exclusion Criteria:

* pregnancy, uncontrolled hemorrhage, terminal heart failure, significant valvular heart disease, documented or suspected acute coronary syndrome, and limitations on the use of inotropes: left ventricle outflow obstruction, systolic anterior motion of the mitral valve.
* incomplete data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Clearances of muscle lactate, and L/P ratio | 3 days
  Clearances of muscle lactate, and L/P ratio were defined as the percentage change in muscle lactate level or L/P ratio compared to baseline (H0) values.

SECONDARY OUTCOMES:
muscle lactate | 3 days
  Interstitial tissue concentration of lactate
muscle pyruvate | 3 days
  Interstitial tissue concentration of pyruvate
muscle glucose | 3 days
  Interstitial tissue concentration of glucose
muscle glycerol | 3 days
  Interstitial tissue concentration of glycerol

CONTACTS AND LOCATIONS:
Overall Officials: zied Hajjej, dr, Principal Investigator — Military hospital
Locations (2):
- Tunisia (2):
  - Military hospital of tunis, Tunis, Mont Fleury
  - Military Hopital of Tunis, Tunis

IPD SHARING:
Plan to Share IPD: No